CLINICAL TRIAL: NCT03783442
Title: A Randomized, Placebo-Controlled, Double-Blind Phase 3 Study to Evaluate the Efficacy and Safety of Tislelizumab (BGB-A317) in Combination With Chemotherapy as First-Line Treatment in Patients With Unresectable, Locally Advanced Recurrent or Metastatic Esophageal Squamous Cell Carcinoma
Brief Title: A Study of Tislelizumab (BGB-A317) in Combination With Chemotherapy as First Line Treatment in Participants With Advanced Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGB-A317-306; 2018-000587-28 (EudraCT Number); CTR20181013 (Other: ChinaDrugTrials); JapicCTI-194741 (Registry Identifier: Japic)
Record Dates: First submitted 2018-12-18; First posted 2018-12-21 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Cisplatin; Oxaliplatin; Fluorouracil; Capecitabine; Paclitaxel; tislelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tislelizumab + Chemotherapy (Experimental): Participants received tislelizumab 200 milligrams (mg) administered intravenously (IV) on Day 1 of each 3-week treatment cycle together with an investigator-chosen chemotherapy doublet until unacceptable toxicity, disease progression or withdrawal for other reasons.
  Chemotherapy options were a platinum agent (cisplatin 60-80 mg/m² intravenously on Day 1 or oxaliplatin 130 mg/m² intravenously on Day 1) combined with a fluoropyrimidine (fluorouracil [750-800 mg/m² intravenously on Days 1-5] or capecitabine [1000 mg/m² orally twice daily on Days 1-14]) or paclitaxel (175 mg/m² intravenously on Day 1).
  Interventions: Drug: Cisplatin; Drug: Oxaliplatin; Drug: Fluorouracil (5-FU); Drug: Capecitabine; Drug: Paclitaxel; Biological: Tislelizumab
- Placebo + Chemotherapy (Active Comparator): Participants received placebo administered IV on Day 1 of each 3-week treatment cycle together with an investigator-chosen chemotherapy doublet until unacceptable toxicity, disease progression or withdrawal for other reasons.
  Chemotherapy options were a platinum agent (cisplatin 60-80 mg/m² intravenously on Day 1 or oxaliplatin 130 mg/m² intravenously on Day 1) combined with a fluoropyrimidine (fluorouracil [750-800 mg/m² intravenously on Days 1-5] or capecitabine [1000 mg/m² orally twice daily on Days 1-14]) or paclitaxel (175 mg/m² intravenously on Day 1).
  Interventions: Drug: Cisplatin; Drug: Oxaliplatin; Drug: Fluorouracil (5-FU); Drug: Capecitabine; Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 60-80 mg/m² administered by intravenous infusion every 3 weeks. Cisplatin was used as the platinum agent in China, Taiwan, and Japan.
Drug: Oxaliplatin — Oxaliplatin 130 mg/m² administered by intravenous infusion every 3 weeks.
Drug: Fluorouracil (5-FU) — Fluorouracil 750-800 mg/m² administered by intravenous infusion on Days 1-5 of each treatment cycle.
Drug: Capecitabine — Capecitabine 1000 mg/m² administered orally twice daily on Days 1-14 of each treatment cycle
Drug: Paclitaxel — Paclitaxel 175 mg/m² administered by intravenous infusion every 3 weeks.
Biological: Tislelizumab — Tislelizumab 200 mg administered by intravenous infusion every 3 weeks.
  Other Names: BGB-A317; TEVIMBRA
  Arms: Tislelizumab + Chemotherapy
Drug: Placebo — Placebo to match tislelizumab administered by intravenous infusion every 3 weeks.
  Arms: Placebo + Chemotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of tislelizumab as first line treatment in combination with chemotherapy in participants with advanced unresectable/metastatic esophageal squamous cell carcinoma (ESCC).

ELIGIBILITY:
Key Inclusion Criteria:

1. Pathologically (histologically) confirmed diagnosis of ESCC
2. Stage IV unresectable ESCC at first diagnosis OR unresectable, locally advanced recurrent or metastatic disease (per American Joint Committee on Cancer 7th Edition), if there is prior neoadjuvant/adjuvant therapy with platinum-based chemotherapy, a treatment-free interval of at least 6 months is required.

Key Exclusion Criteria:

1. Palliative radiation treatment for ESCC within 4 weeks of study treatment initiation
2. Prior systemic therapy for unresectable, locally advanced recurrent or metastatic ESCC
3. Received prior therapies targeting programmed cell death protein-1 (PD-1), programmed cell death protein ligand-1 (PD-L1) or PD-L2
4. Participants with evidence of fistula (either esophageal/bronchial or esophageal/aorta)
5. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage or medical intervention (clinically significant recurrence requiring an additional intervention within 2 weeks of intervention)
6. Evidence of complete esophageal obstruction not amenable to treatment
7. Unintentional weight loss ≥ 5% within one month prior to randomization or Nutritional Risk Index (NRI) < 83.5 per investigator's choice
8. Locally advanced esophageal carcinoma that is resectable or potentially curable with radiation therapy per local investigator.
9. Participants with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers whose HBV DNA is ≥ 500 IU/mL or participants with active hepatitis C virus (HCV)

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 649 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2024-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (124):
- United States (2):
  - Smilow Cancer Hospital At Yale, New Haven, Connecticut
  - Renovatio Clinical, The Woodlands, Texas
- Australia (2):
  - Coffs Harbour Base Hospital, Coffs Harbour, New South Wales
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
- Belgium (6):
  - Institut Jules Bordet, Anderlecht
  - Az Sint Jan Brugge, Bruges
  - Grand Hopital de Charleroi Site Notre Dame, Charleroi
  - UZ GENT, Ghent
  - University Hospitals Leuven, Leuven
  - Chc Montlegia, Liège
- China (42):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Anhui Provincial Cancer Hospital Aka West Branch of Anhui Province Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Fifth Medical Center of Chinese Pla General Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Quanzhou First Affliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospital, Sun Yat Sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Guangdong Province Traditional Chinese Medical Hospitsal, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital, Sun Yat Sen University, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - The Tumor Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Peoples Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital Branch North, Nantong, Jiangsu
  - Affiliated Hospital of Jiangnan University North Campus (Wuxi Fourth Peoples Hospital ), Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Weifang Peoples Hospital, Weifang, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Provincial Peoples Hospital, Taiyuan, Shanxi
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- Fakultni Thomayerova Nemocnice, Prague, Czechia
- France (10):
  - Chru de Brest Hopital Cavale Blanche, Brest
  - Chu Besancon Hopital Jean Minjoz, Doubs
  - Hopital Franco Britannique, LevalloisPerret
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital Saint Antoine Service Dhepato Gastro Enterologie, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Chu Bordeaux Hopital Haut Leveque, Pessac
  - Chu de Poitiers Site de La Mileterie, Poitiers
  - Centre de Lutte Contre Le Cancer Institut de Cancerologie de Louest Rene Gauducheau, SaintHerblain
- Germany (3):
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Slk Kliniken Heilbronn Gmbh Klinik Fur Radiologie, Minimalinvasive Therapien Und Nuklearmedizin, Heilbronn
  - Universitares Krebszentrum Leipzig, Leipzig
- Italy (5):
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori Irst, Meldola
  - Istituto Europeo Di Oncologia, Milan
  - Istituto Nazionale Tumori Fondazione G Pascale, Napoli
  - Iov Istituto Oncologico Veneto Irccs, Padua
  - Azienda Ospedaliera Universitaria Delle Marche, Torrette
- Japan (15):
  - Akita University Hospital, Akitashi, Akita
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Nho Kyushu Cancer Center, Fukuoka, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuokacity, Fukuoka
  - Hyogo Cancer Center, AkashiShi, Hyōgo
  - Johas Kansai Rosai Hospital, Amagasakishi, Hyōgo
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - University Hospital, Kyoto Prefectural Univ of Medicine, KyotoShi, Kyoto
  - Osaka International Cancer Institute, OsakaShi, Osaka
  - The University of Osaka Hospital, Suitashi, Osaka
  - Saitama Cancer Center, Kitaadachigun, Saitama
  - National Cancer Center Hospital, ChuoKu, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - Kumamoto University Hospital, Kumamoto
  - Niigata Cancer Center Hospital, Niigata
- Poland (4):
  - Szpital Specjalist W Brzozowie,Podkarpacki Osrodek Onkologiczny, Brzozów
  - Szpital Wojewodzki Im Mikoaja Kopernika W Koszalinie, Koszalin
  - Spzoz Mswia Z Warminsko Mazurskim Centrum Onkologii, Olsztyn
  - Narodowy Instytut Onkologii Im Marii Skodowskiej Curie Pastwowy Instytut Badawczy, Warsaw
- Romania (4):
  - Institutul Oncologic Prof Dr Ion Chiricuta Cluj Napoca, ClujNapoca
  - Medisprof Cancer Center, ClujNapoca
  - Radiotherapy Center Cluj, ClujNapoca
  - Sc Centrul de Oncologie Sf Nectarie Srl, Craiova
- Russia (7):
  - Arkhangelsk Regional Clinical Oncological Dispensary, Arkhangelsk, Arkhangelskaya oblast
  - Rbih Ivanovo Regional Oncological Dispensary, Ivanovo, Ivanovo Oblast
  - State Budget Healthcare Institution Leningrad Regional Clinical Oncologic Dispensary, Kuzmolovsky, Leningradskaya Oblast'
  - Orenburg Regional Clinical Oncology Center, Orenburg, Orenburg Oblast
  - Rostov State Medical University, RostovonDon, Rostov Oblast
  - Pavlov First Saint Petersburg State Medical University, SaintPetersburg, Sankt-Peterburg
  - Fsbi National Medical Research Center For Oncology Na Nn Petrov of the Moh of the Rf, SaintPetersburg
- South Korea (10):
  - Keimyung University Dongsan Hospital, Dalseogu, Daegu Gwang'yeogsi
  - Cha Bundang Medical Center, Cha University, BundangGu SeongnamSi, Gyeonggi-do
  - Seoul National University Bundang Hospital, BundangGu SeongnamSi, Gyeonggi-do
  - Gachon University Gil Medical Center, NamdongGu, Incheon Gwang'yeogsi
  - Chonnam National University Hwasun Hospital, HwasunGun, Jeollanam-do
  - Smg Snu Boramae Medical Center, DongjakGu, Seoul Teugbyeolsi
  - Korea University Guro Hospital, GuroGu, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St Marys Hospital, SeochoGu, Seoul Teugbyeolsi
  - Samsung Medical Center Hematology Oncology, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, SongpaGu, Seoul Teugbyeolsi
- Spain (7):
  - Hospital Universitario Vall Dhebron, Barcelona
  - Institut Catala Doncologia, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (4):
  - Chiayi Chang Gung Memorial Hospital, Chiayi City
  - Chi Mei Hospital Liouying, Liuying Dist
  - China Medical University Hospital, North Dist
  - Chi Mei Medical Center, Yongkang Dist
- United Kingdom (2):
  - The Christie Hospital, Greater Manchester
  - Guys and St Thomas Hospital Nhs Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/

REFERENCES:
- [Result] Xu J, Kato K, Raymond E, Hubner RA, Shu Y, Pan Y, Park SR, Ping L, Jiang Y, Zhang J, Wu X, Yao Y, Shen L, Kojima T, Gotovkin E, Ishihara R, Wyrwicz L, Van Cutsem E, Jimenez-Fonseca P, Lin CY, Wang L, Shi J, Li L, Yoon HH. Tislelizumab plus chemotherapy versus placebo plus chemotherapy as first-line treatment for advanced or metastatic oesophageal squamous cell carcinoma (RATIONALE-306): a global, randomised, placebo-controlled, phase 3 study. Lancet Oncol. 2023 May;24(5):483-495. doi: 10.1016/S1470-2045(23)00108-0. Epub 2023 Apr 17. PMID 37080222
- [Derived] Xu J, Kato K, Hubner R, Park SR, Kojima T, Ishihara R, Wyrwicz L, Van Cutsem E, Jimenez-Fonseca P, Wu H, Wang L, Yan S, Shi J, Kadva A, Yoon HH. First-Line Tislelizumab Plus Chemotherapy for Esophageal Squamous Cell Carcinoma with Programmed Death-Ligand 1 Expression >/= 1%: A Retrospective Analysis of RATIONALE-306. Adv Ther. 2025 May;42(5):2269-2284. doi: 10.1007/s12325-025-03115-9. Epub 2025 Mar 13. PMID 40075024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 162 centers in 16 countries/regions across Asia, Europe, North America, and Oceania.
Pre-assignment Details: Participants were randomly assigned (1:1), using an interactive response technology system, to either tislelizumab plus investigator-chosen chemotherapy or placebo plus investigator-chosen chemotherapy.
  Randomization was stratified by investigator-chosen chemotherapy (platinum plus fluoropyrimidine vs platinum plus paclitaxel), region (Asia [excluding Japan] vs Japan vs other regions), and previous definitive therapy (yes vs no).
Period: Overall Study
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Started | 326 | 323
Treated | 324 | 321
Completed | 0 | 0
Not Completed | 326 | 323
Not completed — Death | 252 | 268
Not completed — Withdrawal by Subject | 19 | 21
Not completed — Lost to Follow-up | 7 | 6
Not completed — Sponsor Ended Study | 48 | 28

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all randomized participants
Groups:
- Tislelizumab + Chemotherapy: Participants received tislelizumab 200 mg administered IV on Day 1 of each 3-week treatment cycle together with an investigator-chosen chemotherapy doublet until unacceptable toxicity, disease progression or withdrawal for other reasons.
- Placebo + Chemotherapy: Participants received placebo administered IV on Day 1 of each 3-week treatment cycle together with an investigator-chosen chemotherapy doublet until unacceptable toxicity, disease progression or withdrawal for other reasons.
- Total: Total of all reporting groups
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy | Total
Number analyzed (Participants) | 326 | 323 | 649
Age, Continuous [Median (Full Range); unit: years] | 64.0 [26 to 84] | 65.0 [40 to 84] | 64.0 [26 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 42 | 86
  Male | 282 | 281 | 563
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 243 | 243 | 486
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 79 | 76 | 155
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Geographic Region [Count of Participants; unit: Participants] — Rest of World includes Europe, North America and Oceania.
  Participants
    Asia (excluding Japan) | 210 | 210 | 420
    Japan | 33 | 33 | 66
    Rest of World | 83 | 80 | 163
Prior Definitive Therapy [Count of Participants; unit: Participants] — A tumor that is localized without distant metastases is treated with definitive therapy with the intention to cure, and may have included chemotherapy, radiotherapy and/or surgery.
  Participants
    Yes | 152 | 150 | 302
    No | 174 | 173 | 347
Investigator Chosen Chemotherapy [Count of Participants; unit: Participants]
  Platinum with Fluoropyrimidine | 147 | 146 | 293
  Platinum with Paclitaxel | 179 | 177 | 356
Programmed Cell Death Protein Ligand-1 (PD-L1) Expression [Count of Participants; unit: Participants] — PD-L1 is a protein found on some normal cells and in higher-than-normal amounts on certain cancer cells that can block the immune system from attacking cancer cells.
  PD-L1 expression was assessed by a central laboratory using the tumor area positivity (TAP) score, defined as total percentage of tumor area (tumor and any desmoplastic stroma) covered by tumor cells with PD-L1 membrane staining (any intensity), and tumor associated immune cells with PD-L1 staining (any intensity), visually estimated by pathologists using the Ventana PD-L1 (SP263) assay.
  Participants
    PD-L1 Score ≥ 10% | 116 | 107 | 223
    PD-L1 Score < 10% | 151 | 168 | 319
    Unknown | 59 | 48 | 107

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of randomization until the date of death due to any cause. Median OS was estimated using the Kaplan-Meier method.
  Primary analysis (data cut-off date of 28 February 2022) was the pre-defined analysis at which the primary endpoint was tested for superiority.
Time Frame: From randomization to the primary analysis cutoff date of 28 February 2022; maximum time on follow-up was 3 years and 2 months.
Population: The ITT analysis set included all randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 326 | 323
months | 17.2 [15.8 to 20.1] | 10.6 [9.3 to 12.1]
Statistical Analysis 1: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Test type: Superiority; p < 0.0001, Stratified Log-rank Test; One-sided p-value estimated from log rank test stratified by pooled geographic region, prior definitive therapy and Investigator chemotherapy choice; Stratified Hazard Ratio = 0.66, 95% CI 2-sided [0.54 to 0.80] — Stratified Hazard ratio was based on Cox regression model including treatment arm as a covariate and stratified by pooled geographic region (Asia vs. Rest of World), prior definitive therapy and Investigator choice of chemotherapy as strata

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival is defined as the time from the date of randomization to the date of first documentation of disease progression assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, or death, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method.
  Progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, and an absolute increase of at least 5 mm, or unequivocal progression of existing nontarget lesions, or the appearance of 1 or more new lesions.
  Primary analysis (data cut-off date of 28 February 2022) was the pre-defined analysis at which the primary endpoint was tested for superiority. Testing for all secondary efficacy endpoints was conducted at the time of the primary analysis.
Time Frame: as for outcome 1
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 326 | 323
months | 7.3 [6.9 to 8.3] | 5.6 [4.9 to 6.0]
Statistical Analysis 1: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Test type: Superiority; p < 0.0001, Stratified Log-rank test; [statistical method as in outcome 1, analysis 1]; Stratified Hazard Ratio = 0.62, 95% CI 2-sided [0.52 to 0.75] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants whose best overall response (BOR) was complete response (CR) or partial response (PR) assessed by the investigator per RECIST v1.1. Tumor assessments included computed tomography (CT) scans or magnetic resonance imaging (MRI), with preference for CT, of the neck, chest, and abdomen.
  CR: Disappearance of all target and nontarget lesions with no new lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm.
  PR: Disappearance of all target lesions with persistence of 1 or more nontarget lesion(s), no new lesions, and/or maintenance of tumor marker level above the normal limits, or, at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Testing for all secondary efficacy endpoints was conducted at the time of the primary analysis (data cutoff date of 28 February 2022).
Time Frame: Response was assessed every 6 weeks for the first 48 weeks, then every 9 weeks thereafter; up to the primary analysis cutoff date of 28 February 2022; maximum time on follow-up was 3 years and 2 months.
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 326 | 323
percentage of participants | 63.5 [58.0 to 68.7] | 42.4 [37.0 to 48.0]
Statistical Analysis 1: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Two-sided Cochran-Mantel-Haenszel test was stratified by pooled geographic region, prior definitive therapy, and Investigator choice of chemotherapy; Odds Ratio (OR) = 2.38, 95% CI 2-sided [1.73 to 3.27] — Odds ratio was calculated using the Cochran-Mantel-Haenszel method, stratified by pooled geographic region, prior definitive therapy, and Investigator choice of chemotherapy

4. Secondary Outcome: Overall Survival (OS) in Participants With a PD-L1 Score ≥ 10%
Description: OS is defined as the time from the date of randomization until the date of death due to any cause. Median OS was estimated using the Kaplan-Meier method.
  Primary analysis (data cut-off date of 28 February 2022) was the pre-defined analysis at which the primary endpoint was tested for superiority. Testing for all secondary efficacy endpoints was conducted at the time of the primary analysis.
Time Frame: as for outcome 1
Population: ITT Analysis Set participants with PD-L1 score ≥ 10%
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 116 | 107
months | 16.6 [15.3 to 24.4] | 10.0 [8.6 to 13.3]
Statistical Analysis 1: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Test type: Superiority; p = 0.0029, Stratified Log-rank test; [statistical method as in outcome 1, analysis 1]; Stratified Hazard Ratio = 0.62, 95% CI 2-sided [0.44 to 0.87] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the first determination of an objective response until the first documentation of progression assessed by the investigator per RECIST v1.1 or death, whichever occurred first. Median DOR was estimated using the Kaplan-Meier method.
  Primary analysis (data cut-off date of 28 February 2022) was the pre-defined analysis at which the primary endpoint was tested for superiority. Testing for all secondary efficacy endpoints was conducted at the time of the primary analysis.
Time Frame: as for outcome 1
Population: Participants in the ITT Analysis Set with an objective response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 207 | 137
months | 7.1 [6.1 to 8.1] | 5.7 [4.4 to 7.1]

6. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Oesophageal Cancer 18 Question Module (QLQ-OES18) Dysphagia, Eating, Reflux, Pain, and Index Scores
Description: The EORTC-QLQ-OES18 is the specific esophageal symptoms module of the QLQ-C30. QLQ-OES18 is comprised of 18 questions grouped into 4 multi-item subscales: Dysphagia (3 items), Eating (4 items), Reflux (2 items), and Pain (3 items) and 6 single item subscales (trouble swallowing saliva, choking, dry mouth, taste, coughing, and talking). Participants indicate the extent to which they have experienced symptoms on a scale from 1 (Not at all) to 4 (Very much). Scores are calculated as the average of the items that contribute to the scale, then transformed to a scale from 0 to 100. The OES18 index score is calculated as the average of the 4 multi-item subscales and 6 single-item subscales. Higher scores indicate a higher level of symptomatology or problems.
Time Frame: Baseline, Cycle 6 (Week 15)
Population: Participants in the ITT Analysis Set who completed the EORTC QLQ-OES18 at Baseline and at least one post-baseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 310 | 309
score on a scale
  Dysphagia | -0.5 [-4.7 to 3.7] | -4.9 [-9.4 to -0.5]
  Eating | -0.9 [-3.1 to 1.3] | -1.5 [-3.8 to 0.9]
  Reflux | -1.3 [-3.2 to 0.7] | 0.2 [-1.9 to 2.2]
  Pain | -5.2 [-6.7 to -3.7] | -3.3 [-4.9 to -1.8]
  Index Score | -1.0 [-2.2 to 0.3] | -0.6 [-1.9 to 0.7]
Statistical Analysis 1: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in EORTC QLQ-OES18 Dysphagia Score at Cycle 6; Test type: Superiority; p = 0.1372, Mixed Models Analysis; Two-sided p-value estimated from a mixed effect model; Least Squares (LS) Mean Difference = 4.4, 95% CI 2-sided [-1.4 to 10.3] — Based on a mixed effect model analysis with QLQ-OES18 scores until cycle 18 as the response variable, and treatment by study visit interaction, Baseline mean score, and randomization stratification factors as covariates
Statistical Analysis 2: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in EORTC QLQ-OES18 Eating Score at Cycle 6; Test type: Superiority; p = 0.7130, Mixed Models Analysis; Two-sided p-value estimated from a mixed effect model; LS Mean Difference = 0.6, 95% CI 2-sided [-2.5 to 3.7] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in EORTC QLQ-OES18 Reflux Score at Cycle 6; Test type: Superiority; p = 0.3001, Mixed Models Analysis; Two-sided p-value estimated from a mixed effect model; LS Mean Difference = -1.4, 95% CI 2-sided [-4.1 to 1.3] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in EORTC QLQ-OES18 Pain Score at Cycle 6; Test type: Other; LS Mean Difference = -1.9, 95% CI 2-sided [-3.9 to 0.2] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in EORTC QLQ-OES18 Index Score at Cycle 6; Test type: Other; LS Mean Difference = -0.4, 95% CI 2-sided [-2.1 to 1.4] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Core 30 (QLQ-C30) Global Health Status/Quality of Life (GHS/QoL) and Physical Functioning Scales
Description: The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 = Not at all (best) and 4 = Very Much (worst) and 2 global health quality of life (QOL) questions answered on a 7-point scale where 1 = Very poor and 7 = Excellent. Raw scores are transformed to a 0 to 100 scale via linear transformation. Higher scores in GHS and functional scales indicate better quality of life.
Time Frame: Baseline, Cycle 6 (Week 15)
Population: Participants in the ITT Analysis Set who completed the EORTC QLQ-C30 at Baseline and at least one post-baseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 310 | 309
score on a scale
  Global Health Status/ QOL | -0.3 [-2.3 to 1.8] | -3.6 [-5.8 to -1.4]
  Physical Functioning | -4.8 [-6.6 to -3.0] | -7.3 [-9.2 to -5.4]
Statistical Analysis 1: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in Global Health Status/QoL at Cycle 6; Test type: Other; LS Mean Difference = 3.3, 95% CI 2-sided [0.4 to 6.2] — Based on a mixed effect model analysis, with QLQ-C30 scores until cycle 18 as the response variable, and treatment by study visit interaction, Baseline mean score, and randomization stratification factors as covariates
Statistical Analysis 2: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Analysis of Change from Baseline in Physical Functioning at Cycle 6; Test type: Other; LS Mean Difference = 2.6, 95% CI 2-sided [0.0 to 5.1] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Fatigue Scale
Description: The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 = Not at all (best) and 4 = Very Much (worst) and 2 global health quality of life (QOL) questions answered on a 7-point scale where 1 = Very poor and 7 = Excellent. Raw scores are transformed to a 0 to 100 scale via linear transformation. The fatigue symptom scale includes 3 items and ranges from 0 to 100, where higher scores indicate a higher level of symptoms.
Time Frame: Baseline, Cycle 6 (Week 15)
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 310 | 309
score on a scale | 8.0 [5.7 to 10.4] | 9.4 [6.9 to 11.9]
Statistical Analysis 1: Comparison: Tislelizumab + Chemotherapy vs Placebo + Chemotherapy; Test type: Other; LS Mean Difference = -1.4, 95% CI 2-sided [-4.7 to 1.9] — Based on a mixed effect model analysis with QLQ-C30 scores until cycle 18 as the response variable, and treatment by study visit interaction, Baseline mean score, and randomization stratification factors as covariates

9. Secondary Outcome: Change From Baseline in European Quality of Life 5-Dimension 5-Level (EQ-5D-5L) Visual Analog Scale (VAS)
Description: The EQ-5D-5L measures health outcomes using a VAS to record a participant's self-rated health on a scale from 0 to 100, where 100 is 'the best health you can imagine' and 0 is 'the worst health you can imagine.' A higher score indicates better health outcomes.
Time Frame: Baseline, Cycle 6 (Week 15)
Population: Participants in the ITT Analysis Set with EQ-5D-5L measurement at both Baseline and Cycle 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 221 | 196
score on a scale | -1.1 (15.82) | -3.1 (14.01)

10. Secondary Outcome: Number of Participants Experiencing Treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drugs, whether related to study drugs or not.
  An SAE is any untoward medical occurrence that, at any dose met any of the following criteria:
  * Resulted in death
  * Was life-threatening
  * Required hospitalization or prolongation of existing hospitalization
  * Resulted in disability/incapacity
  * Was a congenital anomaly/birth defect
  * Was considered a significant medical AE by the Investigator based on medical judgement.
Time Frame: From first dose of study drug up to 30 days after last dose; maximum time on treatment was 63.5 months.
Population: Safety analysis set included all participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
Number analyzed (Participants) | 324 | 321
Participants
  Treatment-emergent adverse event | 323 | 319
  Serious adverse events | 160 | 128

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from randomization until the end of study, maximum time on study was 63.6 months. Adverse events were assessed from first dose of study drug to 30 days after last dose, maximum time on treatment was 63.5 months.
Description: All-cause mortality was assessed in all randomized participants; adverse events were assessed in all participants who received at least 1 dose of study drug.
Arm/Group | Tislelizumab + Chemotherapy | Placebo + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 252/326 | 268/323
Serious Adverse Events (participants affected / at risk) | 160/324 | 128/321
Other Adverse Events (participants affected / at risk) | 321/324 | 314/321
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab + Chemotherapy (N=324) | Placebo + Chemotherapy (N=321)
Anaemia (Blood and lymphatic system disorders) | 6 (8) | 6 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 5 (5)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 4 (5)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 7 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (2)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 3 (3) | 0 (0)
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 3 (3) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 17 (17) | 8 (8)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 3 (5)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (3)
Oesophageal dysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 3 (3) | 3 (3)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Oesophageal obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 7 (7) | 2 (2)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 5 (6) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (8) | 5 (5)
Accidental death (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (3) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 3 (3)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 4 (4)
Fatigue (General disorders) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 6 (6) | 4 (4)
Malaise (General disorders) | 5 (5) | 3 (3)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (6) | 1 (1)
Sudden death (General disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (2)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Anaphylactic shock (Immune system disorders) | 2 (2) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium colitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic infection (Infections and infestations) | 0 (0) | 1 (2)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 19 (21) | 23 (23)
Post procedural pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 2 (2) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 2 (2)
Septic shock (Infections and infestations) | 3 (3) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Urethritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Oropharyngeal stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Unintentional medical device removal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (5) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 3 (3)
Prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 2 (3) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (7) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Immune-mediated arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Malignant spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mutism (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular dysfunction (Renal and urinary disorders) | 0 (0) | 1 (1)
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (4)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab + Chemotherapy (N=324) | Placebo + Chemotherapy (N=321)
Anaemia (Blood and lymphatic system disorders) | 193 (343) | 180 (322)
Coagulopathy (Blood and lymphatic system disorders) | 13 (15) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 34 (86) | 28 (87)
Neutropenia (Blood and lymphatic system disorders) | 54 (122) | 45 (148)
Thrombocytopenia (Blood and lymphatic system disorders) | 29 (43) | 24 (36)
Hypothyroidism (Endocrine disorders) | 33 (35) | 15 (21)
Abdominal distension (Gastrointestinal disorders) | 17 (29) | 14 (19)
Abdominal pain (Gastrointestinal disorders) | 25 (26) | 13 (17)
Abdominal pain upper (Gastrointestinal disorders) | 15 (19) | 13 (20)
Constipation (Gastrointestinal disorders) | 102 (141) | 101 (130)
Diarrhoea (Gastrointestinal disorders) | 88 (124) | 76 (118)
Dyspepsia (Gastrointestinal disorders) | 13 (21) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 32 (41) | 29 (30)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 23 (26) | 15 (17)
Nausea (Gastrointestinal disorders) | 122 (203) | 136 (229)
Stomatitis (Gastrointestinal disorders) | 60 (113) | 48 (67)
Vomiting (Gastrointestinal disorders) | 68 (112) | 86 (145)
Asthenia (General disorders) | 42 (55) | 46 (55)
Chest discomfort (General disorders) | 13 (14) | 4 (4)
Fatigue (General disorders) | 64 (84) | 55 (77)
Malaise (General disorders) | 40 (77) | 51 (70)
Non-cardiac chest pain (General disorders) | 11 (16) | 11 (14)
Oedema peripheral (General disorders) | 14 (17) | 12 (30)
Pyrexia (General disorders) | 54 (80) | 38 (46)
Conjunctivitis (Infections and infestations) | 10 (11) | 3 (3)
Nasopharyngitis (Infections and infestations) | 10 (11) | 6 (6)
Pneumonia (Infections and infestations) | 26 (28) | 14 (15)
Upper respiratory tract infection (Infections and infestations) | 29 (36) | 17 (19)
Alanine aminotransferase increased (Investigations) | 49 (76) | 42 (61)
Amylase increased (Investigations) | 22 (43) | 19 (27)
Aspartate aminotransferase increased (Investigations) | 51 (86) | 37 (57)
Blood alkaline phosphatase increased (Investigations) | 18 (28) | 15 (20)
Blood bilirubin increased (Investigations) | 27 (40) | 27 (44)
Blood creatine phosphokinase increased (Investigations) | 13 (26) | 8 (16)
Blood creatinine increased (Investigations) | 47 (83) | 30 (73)
Blood lactate dehydrogenase increased (Investigations) | 18 (24) | 9 (13)
Blood urea increased (Investigations) | 24 (51) | 16 (32)
Gamma-glutamyltransferase increased (Investigations) | 16 (23) | 17 (21)
Lipase increased (Investigations) | 18 (24) | 17 (25)
Lymphocyte count decreased (Investigations) | 23 (57) | 28 (65)
Neutrophil count decreased (Investigations) | 153 (497) | 155 (486)
Platelet count decreased (Investigations) | 62 (121) | 55 (111)
Weight decreased (Investigations) | 97 (125) | 91 (112)
Weight increased (Investigations) | 29 (39) | 13 (13)
White blood cell count decreased (Investigations) | 143 (487) | 157 (520)
Decreased appetite (Metabolism and nutrition disorders) | 142 (205) | 124 (195)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 13 (27) | 7 (21)
Hyperglycaemia (Metabolism and nutrition disorders) | 33 (48) | 26 (35)
Hyperkalaemia (Metabolism and nutrition disorders) | 22 (33) | 17 (33)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 16 (37) | 13 (28)
Hyperuricaemia (Metabolism and nutrition disorders) | 27 (78) | 25 (61)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 75 (157) | 60 (115)
Hypocalcaemia (Metabolism and nutrition disorders) | 20 (28) | 17 (28)
Hypochloraemia (Metabolism and nutrition disorders) | 37 (64) | 31 (52)
Hypokalaemia (Metabolism and nutrition disorders) | 64 (105) | 54 (83)
Hypomagnesaemia (Metabolism and nutrition disorders) | 31 (68) | 29 (41)
Hyponatraemia (Metabolism and nutrition disorders) | 73 (129) | 58 (99)
Hypophosphataemia (Metabolism and nutrition disorders) | 16 (22) | 15 (24)
Hypoproteinaemia (Metabolism and nutrition disorders) | 14 (18) | 12 (21)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (37) | 32 (45)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (26) | 20 (25)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 10 (12) | 7 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 28 (42) | 22 (29)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 (37) | 29 (36)
Dizziness (Nervous system disorders) | 16 (18) | 17 (23)
Dysgeusia (Nervous system disorders) | 12 (14) | 11 (13)
Headache (Nervous system disorders) | 18 (22) | 16 (16)
Hypoaesthesia (Nervous system disorders) | 34 (35) | 40 (44)
Neurotoxicity (Nervous system disorders) | 16 (19) | 11 (12)
Paraesthesia (Nervous system disorders) | 15 (17) | 8 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 74 (82) | 62 (81)
Insomnia (Psychiatric disorders) | 30 (36) | 26 (34)
Cough (Respiratory, thoracic and mediastinal disorders) | 51 (62) | 38 (45)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 11 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (24) | 14 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 23 (35) | 28 (47)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 6 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 25 (27) | 18 (22)
Alopecia (Skin and subcutaneous tissue disorders) | 61 (61) | 63 (63)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (16) | 7 (7)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 14 (17) | 14 (16)
Pruritus (Skin and subcutaneous tissue disorders) | 45 (56) | 21 (27)
Rash (Skin and subcutaneous tissue disorders) | 38 (53) | 24 (30)
Hypertension (Vascular disorders) | 21 (29) | 17 (24)
Hypotension (Vascular disorders) | 14 (19) | 5 (5)
Phlebitis (Vascular disorders) | 7 (7) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT03783442/Prot_002.pdf
  • Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/42/NCT03783442/SAP_001.pdf